CLINICAL TRIAL: NCT04169321
Title: First in Human Safety of [68Ga]-NOTA-hGZP- PET Imaging in Subjects Receiving Checkpoint Inhibitor Immunotherapy
Brief Title: Granzyme B PET Imaging Drug as a Predictor of Immunotherapy Response to Checkpoint Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytosite Biopharma Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other); University of Alabama at Birmingham (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-hGZP-101.12
Record Dates: First submitted 2019-11-04; First posted 2019-11-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Unspecified, Adult; Lymphoma
Keywords: cancer immunotherapy; biomarkers, tumor; positron-emission tomography; Granzymes
MeSH Terms: conditions — Lymphoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: Multiple center, open label, non-randomized, single dose study, in subjects with cancer undergoing or treatment with a checkpoint inhibitor either as a monotherapy or in combination. subjects. Eligible subjects will receive an injection of [68Ga]-NOTA-hGZP pre checkpoint inhibitor administration and a second dose between 5 and 42 days post initial checkpoint inhibitor administration. Upon dosing each subject will undergo PET scans at 40, 60 and 90 minutes post dosing. The images will be analyzed for the distribution of radioactivity. Subjects will be followed for adverse events for approximately 4-6 hours post injection or until pembrolizumab injection plus a follow up phone call to assess adverse events 1-3 days after injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): All participants will receive a mass dose of 40 μg or less of [68Ga]-NOTA-hGZP (radioactivity dose of 3 mCi to 8 mCi) and have a PET and CT scan.
  Interventions: Drug: Single Arm

INTERVENTIONS:
Drug: Single Arm — [68Ga]-NOTA-hGZP is a PET imaging agent.
  Other Names: [68Ga]-NOTA-hGZP; CSB-111

SUMMARY:
First in Human Safety of [68Ga]-NOTA-hGZP PET Imaging in subjects with cancer undergoing treatment with a checkpoint inhibitor either as a monotherapy of in combination I-O therapy

DETAILED DESCRIPTION:
This is a first in human research study (Phase I clinical trial) to test the safety and effectiveness of a new radioactive PET imaging drug and biomarker [68Ga]-NOTA-hGZP. It is a multi-center, open label, non-randomized, two dose study to evaluate the safety of [68Ga]-NOTA-hGZP and the ability to predict the clinical response to checkpoint inhibitor therapy within 2 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age and older.
2. Subjects with proven metastatic cancer that is going to be treated with one or more checkpoint inhibitors under the licensed indications for the cancer type. Checkpoint inhibitors include PD-1, PD-L1, CTLA-4 and LAG-3 inhibitors.
3. Subjects must have at least one lesion ≥ 15 mm in diameter or with two lesions both ≥ 15mm in diameter, when an optional biopsy is planned. Lesion measurements are taken from a diagnostic quality CT or MR image.
4. ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
5. Life expectancy of greater than 6 months.
6. Males and females willing to use adequate contraception prior to study and during study participation.
7. If female, not of childbearing potential or negative pregnancy test prior to radiotracer injection.
8. Willing and able to understand and sign a written informed consent document.
9. Willing and able to undergo all study procedures.
10. Cohort 3 only: have archival lesion tissue available within 90 days of enrollment either from biopsy or surgery.

Exclusion Criteria:

1. Participants for whom adverse events due to agents administered more than 4 weeks earlier have not resolved to Grade 1 or less.
2. Has not received nor is expected to receive an investigational compound within 90 days prior to [68Ga]-NOTA-hGZP PET imaging. This includes checkpoint inhibitors that are not approved by the US FDA for the indications in this protocol.
3. Subjects who have received a prior checkpoint inhibitor.
4. Any acute or chronic inflammatory disease or medical conditions that in the investigator's opinion may interfere with the study procedures or the interpretation of the study results such as infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
5. Known brain metastases.
6. History of allergic reactions to compounds of similar chemical or biologic composition to [68Ga]-NOTA-hGZP or pembrolizumab.
7. If female, nursing.
8. Current treatment with systemic steroids, or immunosuppressive agents. Participants with a condition requiring systemic treatment with either corticosteroids (< 10 mg daily prednisone equivalent) inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
9. Subjects who have exclusion criteria that would prevent them from receiving a CT scan.
10. Laboratory values

    1. Leukocytes < 3000/mcL
    2. Absolute neutrophil count < 1500 mcL
    3. Platelets < 100,000 mCL
    4. Total bilirubin > 1.5 x ULN
    5. AST/ALT > 2.5 x ULN
    6. Albumin < 2 g/dL
    7. Alkaline phosphatase > 2.5 ULN
    8. eGRF eGFR < 45 mL/min/1.73 m2

Patients who are stable but have values outside the specified ranges may be included with approval of the study medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically meaningful changes in physical examination findings, vital signs or blood chemistry | up to 4 to 6 hours post-injection
  Clinically significant changes from baseline in physical examination findings
  Clinically significant changes from baseline to follow-up analysis in systolic and diastolic blood pressure (mmHg)
  Clinically significant changes from baseline to follow-up analysis in heart rate (beats per minute)
  Clinically significant changes in respiration rate.
  Clinically significant changes from baseline to follow-up analysis in blood chemistry for:
  1. Leukocytes (/mcL),
  2. Absolute neutrophil count (mcL)
  3. Platelets (/mcL)
  4. Total bilirubin (mg/d)
  5. AST/ALT (unitless)
  6. Albumin (g/dL)
  7. Alkaline phosphatase (IU/L)
  8. eGRF (mL/min/1.73 m2)
Number of participants with changes in ECG | up to 4 to 6 hours post-injection
  Clinically significant changes from baseline to follow-up analysis in ECG change in QT (ms) Quantification of [68Ga]-NOTA-hGZP PET accumulation at tumor site in subjects after treatment with checkpoint inhibitor therapy as determined by region of interest analysis (SUVmean).
Number of participants with treatment-related Adverse Events (AEs) | Between time of injection and 3 days post injection
  The absolute number of participants with AEs according to CTCAE 5.0

SECONDARY OUTCOMES:
Evaluation of the accumulation of [68Ga]-NOTA-hGZP in tumor foci in participants receiving checkpoint inhibitor therapy (absolute number of avid lesions per subject) | up to one-hour post injection
  Identification by the central reader of the number of avid lesions observed in each subject and the number of subjects with avid lesions seen on the PET images
Quantification of accumulation of [68Ga]-NOTA-hGZP in tumor foci in participants receiving checkpoint inhibitor therapy. | up to one-hour post injection
  To be determined by region of interest analysis the mean standardized uptake value (SUVmean) (SUV does not have any units)
Evaluate the correlation of [68Ga]-NOTA-hGZP accumulation in tumor foci to 6-month outcome. | 6 months
  Compare quantified [68Ga]-NOTA-hGZP uptake to participant treatment response in individual lesions as assessed at 6-month clinical follow-up and/or CT assessments.
  The number of lesions that were avid and the lesions that showed a decrease in size compared to those which increased in size.
Correlate uptake of [68Ga]-NOTA-hGZP tracer and granzyme B expression as assessed on optional excisional biopsy when available (melanoma only). | up to one-hour post injection
  Compare granzyme B protein quantification from biopsied tissue to the [68Ga]-NOTA-hGZP PET uptake acquired at the same location.

CONTACTS AND LOCATIONS:
Overall Officials: Colin G Miller, PhD, Study Director — CytoSite Bio Inc.
Locations (3):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Massachusetts General Hospital, Boston, Massachusetts
- Chang-Gung Memorial Hospital, Taoyuan, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No